CLINICAL TRIAL: NCT05195190
Title: Validity, Reliability and Minimum Detectable Changes of 2-Minute Walk , Timed Up and Go, Sit and Stand Test in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, Assistant professor, Acibadem University
Other Study IDs: ATADEK 2021 -21/19
Record Dates: First submitted 2021-12-14; First posted 2022-01-18 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical test — The 2 minutes walking test, the time up and go test and the 30 second sit and stand test will be applied to the patients in order. Each test will be repeated 2 times after the familiarization test and the average of the tests will be taken. There will be a 10-minute rest period between tests. For the re-test, the tests will be repeated after the patients are given a rest period of 2 hour. Testing will be conducted by a single therapist with at least 5 years of experience blinded to the study.

SUMMARY:
Prostate cancer is a type of cancer that can occur in men, especially in the fifth and sixth decades of their lives, and various side effects occur depending on the treatments applied in the diagnosed patients. The treatments applied and the decreased level of physical activity also cause a decrease in the quality of life. Recent studies have focused on treatment-related side effects. Before treatment planning, there is a need for clinically validated clinical evaluations specific to prostate cancer patients in order to determine the current status of the patients or to measure the effectiveness of the treatment applied. In addition, tests with a minimal detectable amount of change will be guiding in order to understand that the effectiveness of the applied treatment is significant. The aim of our study is to investigate the validity, reliability and minimal detectable changes of the two-minute walk, sit up and time up and go tests validated in different disease groups for patients with prostate cancer.

DETAILED DESCRIPTION:
Performance-based outcome measures are gaining importance in terms of patients' health care. These tests are not specific for any disease or extremity. They are specific tests for walking and getting up from a chair. They evaluate what an individual can do rather than what they perceive the individual can do. Performance measurement tests have a higher level of evidence than just self-reported evaluations.

Time up and go test, two-minute walk test, sit and stand test are the most frequently used tests in the clinic to evaluate functionality. The short duration of the tests and the fact that they do not require equipment provide advantages in the clinical setting.

In the current literature, the validity and reliability of the Time up and go, two-minute walk and sit-up test in elderly prostate cancer patients has not been established. The aim of our study is to investigate the validity and reliability of these tests in elderly prostate cancer patients and to determine their minimum detectable change. Our second aim is to investigate the relationship of these tests we evaluated with the Nottingham Health Profile questionnaire, which evaluates health-related quality of life in elderly cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving or continuing Androgen deprivation therapy for at least 3 months
* Diagnosed with non-metastatic prostate cancer
* In the process of radiotherapy or chemoradiotherapy
* Able to walk without assistive device
* Patients over 55 years of age

Exclusion Criteria:

* Diagnosed with metastatic prostate cancer
* Uncontrollable cardiovascular disease Uncontrollable insulin due to diabetes Individuals with neuromuscular, metabolic disease that may effect physical tests

Ages: 55 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Volunteer patients between 55 and 75 years of age with non metastatic prostate cancer will be recruited by simple randomization.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
2 minute walk test -2MWT | 2 hours
  You will be instructed to "walk at a comfortable, usual pace". There will be two attempts for application trial and registration. Practice trial will be used to minimize any potential learning impact. After resting for at least 10 minutes between trials, the distance traveled in 2 minutes will be recorded as 2MWT. The average of both tests will be taken
Time Up and Go Test | 2 hours
  It is the time measured when an individual is standing, walking 3 m straight, returning to the chair, and sitting. In the study, the you will sit comfortably in a chair without back support and arm support. The time for the test will begin as soon as you get up from the chair and will end after you sit in the chair. If the test is less than 10 seconds, it indicates functional independence, and if it is over 30 seconds, it indicates functional dependence.
Sit and Stand Test | 2 hours
  It is used to measure lower extremity strength and evaluate physical capacity. For this study, you will be asked to get up and sit as much as they can within 30 seconds from a chair with a standard 17-inch sitting height and back support.

SECONDARY OUTCOMES:
Nottingham Health Profile -NHP | through study completion, an average of 6 months
  The Turkish version of the NHP will be used to assess health-related quality of life. NHP is a general quality of life questionnaire that measures the perceived health problems of the individual and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items and evaluates 6 sub-dimensions related to health status. Energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). Questions are answered with yes or no. Each section is scored between 0-100. 0 indicates best health, 100 indicates worst health

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Mehmet Ali Aydınlar University, Istanbul, Turkey (Türkiye)